CLINICAL TRIAL: NCT01948180
Title: A Phase 2 Single Arm Study to Investigate the Efficacy of Autologous EBV-specific T-cells for the Treatment of Patients With Aggressive EBV Positive Extranodal NK/T-cell Lymphoma (ENKTCL)
Brief Title: Cellular Immunotherapy Treatment Antigen-Directed for EBV Lymphoma
Acronym: CITADEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment rate
Sponsor: Cell Medica Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM-2013-01
Record Dates: First submitted 2013-09-13; First posted 2013-09-23 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Lymphoma, Extranodal NK-T-Cell; EBV
Keywords: NKTCL; T cell; CITADEL; Epstein-Barr Virus; Natural Killer
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- baltaleucel-T (Experimental): Treatment consists of 2 infusions of 2x10E7 cells/m2 given on Days 1 and 15 intravenously via a peripheral or central line over a 1 to 10 minute period.
  Subjects who tolerate the study treatment well and who do not require treatment with an alternative chemotherapeutic agent will be eligible for up to 3 additional infusions of 2x10E7 cells/m2 administered at week 8, month 3 and month 6.
  Interventions: Biological: baltaleucel-T

INTERVENTIONS:
Biological: baltaleucel-T — Autologous EBV-specific T-cells
  Other Names: CMD-003

SUMMARY:
To investigate the efficacy of autologous EBV-specific T-cells for the treatment of patients with aggressive EBV positive extranodal NK/T-cell lymphoma

ELIGIBILITY:
FOR SCREENING PHASE:

Inclusion Criteria:

1. Diagnosis of extranodal NK/T lymphoma, per WHO classification, 4th ed., which must include EBV tumor positivity, measured either by EBV encoded RNA (EBER) or LMP1 immunostaining.
2. a) Active Disease

(1) Clinically suspected or documented relapse/progression, in first or second relapse following at least one cycle of an asparaginase-based chemotherapy regimen OR (2) Initial disease or first or second relapse and unable to tolerate one full cycle of asparaginase-based chemotherapy regimen OR b) High-risk disease (stage III/IV, KPI groups 3-4 or IPI intermediate-high) prior to second CR regardless of previous chemotherapy.

3. Male or female ≥ 18 years of age. 4. Weigh ≥ 35 kg. 5. ECOG performance score 0-2, inclusively. 6. Negative β-hCG test in women of childbearing potential. 7. Able to understand and comply with the requirements of the study and to provide written informed consent.

Exclusion Criteria:

1. CNS lymphoma.
2. NK cell leukemia.
3. Hemophagocytic lymphohistiocytosis.
4. Positive for HIV, hepatitis B, hepatitis C, syphilis or human T Cell leukemia virus (HTLV).
5. Use of systemic corticosteroids >0.5 mg/kg/day within 10 days prior to obtaining 200 mL whole blood starting material.
6. Patient is pregnant or lactating.
7. Active second malignancy.
8. Any prior allogeneic hematopoietic stem cell or solid organ transplant.
9. Asparaginase refractory disease, defined by any one of the following:

   1. Progression at any time during initial asparaginase based chemotherapy and up to 3 months after end of initial asparaginase based chemotherapy, OR
   2. Failure to achieve at least PR with initial asparaginase based chemotherapy.
10. Absolute lymphocyte count (ALC) <400/µL.
11. Any previous autologous EBV specific T cell treatment.
12. Systemic fungal, bacterial, viral or other infection that is not controlled.
13. Third or greater relapse.

FOR TREATMENT PHASE:

Inclusion Criteria:

1. Documented relapse or progression following at least one prior cycle of an asparaginase-containing chemotherapy regimen.
2. Active disease based on any one of the following present at the baseline study visit or within two weeks prior to the baseline study visit:

   1. Imaging (may use local imaging)
   2. Clinical sign(s) including skin lesions consistent with lymphoma, organ dysfunction or organomegaly not attributable to other causes; or other clinical sign(s)
   3. Detectable blood or plasma ENV DNA (may use local laboratory)
3. Completed most recent course of chemotherapy at least 2 weeks prior to first study drug dose.
4. Recovery from acute hematological, hepatic and renal chemotherapy-related toxicities as defined by ≤ Grade 1 according to NCI CTCAE v4.0.
5. Life expectancy ≥ 8 weeks.

Exclusion Criteria:

1. Use of any investigational agents within prior 4 weeks.
2. Radiotherapy within prior 3 weeks.
3. Major surgery within prior 2 weeks.
4. Systemic corticosteroids within 24 hours prior to study drug administration.
5. Evidence of hepatic dysfunction based on serum total bilirubin >3 times upper limit of normal (ULN), or ALT >5 times ULN or AST >5 times ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  Defined as best observed response (complete response or partial response) per Lugano 2014 Disease Response Criteria.

SECONDARY OUTCOMES:
Complete Response Rate | 1 year
Response Duration | 2 years
Time to Response | 1 year
Progression Free Survival | 2 years
Disease Free Survival | 2 years
Overall Survival | 2 years
Adverse Events | 1 year

OTHER OUTCOMES:
Immunological assessment of EBV-specific T-cell activity and phenotyping | 1 year
Monitor levels of plasma and whole blood EBV DNA (viral load) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine; Kurt Gunter, MD, Study Director — Cell Medica
Locations (11):
- United States (5):
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Universitaire Ouest, Paris
  - Centre Hospitalier de Lyon, Pierre-Bénite
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Asan Cancer Center, Seoul
- United Kingdom (2):
  - University College London Hospital, London, UK
  - The Christie Clinic, Manchester, UK

IPD SHARING:
Plan to Share IPD: No